CLINICAL TRIAL: NCT04148872
Title: Mixed Methods Investigation of Chronic Facial Paralysis in Individuals With Synkinesis: Study of Outcomes Before and After Treatment
Brief Title: Mixed Methods Investigation of Chronic Facial Paralysis in Individuals With Synkinesis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2019-0406; A539770 (Other: UW Madison); SMPH/SURGERY/SURGERY*OT (Other: UW Madison); Protocol Version 4/15/2020 (Other: UW Madison)
Record Dates: First submitted 2019-10-30; First posted 2019-11-04 (Actual); Results first posted 2022-09-29 (Actual); Last update posted 2022-09-29 (Actual); Status verified 2022-08

CONDITIONS: Synkinesis
MeSH Terms: conditions — Synkinesis | interventions — Nerve Block; Botulinum Toxins, Type A; incobotulinumtoxinA

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Neuromuscular Retraining Therapy (Active Comparator): Neuromuscular retraining therapy alone for four months, with botulinum toxin injection added during an additional four month period.
  Interventions: Other: Neuromuscular Retraining Therapy (4 months); Other: Neuromuscular Retraining + Chemodenervation
- Chemodenervation (Active Comparator): Ipsilateral chemodenervation with botulinum toxin injections alone for four months (onabotulinumtoxinA/Botox, Allergan or incobotulinumtoxinA/Xeomin, Merz), with neuromuscular retraining therapy added for an additional four months.
  Interventions: Drug: Chemodenervation (4 months); Other: Neuromuscular Retraining + Chemodenervation

INTERVENTIONS:
Other: Neuromuscular Retraining Therapy (4 months) — Neuromuscular retraining is an intervention where facial therapists utilize voluntary input to access improved movement patterns in patients with synkinesis.
  Arms: Neuromuscular Retraining Therapy
Drug: Chemodenervation (4 months) — A neurotoxin that temporarily reduces muscle activity and minimizes the effects of uncoordinated muscle.
  Other Names: onabotulinumtoxin A; Botox; incobotulinumtoxin A; Xeomin
  Arms: Chemodenervation
Other: Neuromuscular Retraining + Chemodenervation — Participants will receive both interventions for the last 4 months of their time on study.

SUMMARY:
This proposal will prospectively assess the social, physical, and emotional recognition function in participants with synkinesis. It will measure the effectiveness of neuromuscular retraining therapy to improve muscle coordination compared to chemodenervation, the more established treatment modality, in a single-blinded, randomized control trial using clinician- and patient-reported outcomes measures. The hypothesis tested is that participants undergoing neuromuscular retraining therapy will achieve greater improvement on clinical outcome measures as compared to participants receiving chemodenervation.

In this clinical trial, 36 participants undergoing treatment for synkinesis will be enrolled into one of two treatment arms: chemodenervation or neuromuscular retraining therapy. Participants can expect to be on study for approximately 8 months.

Participants who enroll in this mixed methods investigation will be recruited from patients of the University of Wisconsin Facial Nerve Clinic and also be enrolled in a another study for assessment [Perception of Emotion Expression in Clinical Populations with Facial Paralysis, IRB approval 2015-0366].

DETAILED DESCRIPTION:
Facial nerve paralysis is a devastating event that in up to 30% of cases may result in chronic weakness and/or the disfiguring condition of synkinesis, a long-lasting muscle discoordination of facial movement caused by aberrant facial nerve regeneration after facial nerve paralysis. This is believed to have a detrimental effect on social interactions, mental health, and quality of life.

Neuromuscular retraining therapy and ipsilateral chemodenervation into discoordinated muscles by injection (onabotulinumtoxinA/Botox, Allergan or incobotulinumtoxinA/Xeomin, Merz) are two common treatments for the abnormal muscle movements found in synkinesis. No study has compared the effectiveness of these treatment modalities for synkinesis. Retrospective data including our series at the University of Wisconsin Facial Nerve Clinic show significant benefit of retraining therapy using clinician- and patient-reported outcome measures. However, the manner in which this therapy may be optimized for use in treatment of the sequelae of facial paralysis is unclear. While literature shows beneficial improvement in outcomes with chemodenervation in prospective studies, no study has explored the effectiveness of physical therapy for synkinesis in a controlled, prospective manner. Further, the efficacy of therapy has not been shown to improve recognition and emotional information interpretation, both thought to be impaired in synkinesis.

This study has 3 specific aims:

AIM 1: Determine the effect of neuromuscular retraining or chemodenervation on clinician-reported and patient-reported outcomes. The primary outcome measure after four and eight months of treatment will be the clinician-reported Sunnybrook Facial Grading System (SFGS) scored on participant videos by blinded reviewers. Further, the investigators seek to measure the efficacy of treatment with existing patient-reported instruments. A correlation of clinician-reported outcome measure changes to changes in patient-reported instruments with treatment will be calculated, including the widely utilized disease specific Synkinesis Assessment Questionnaire (SAQ) and Facial Clinimetric Evaluation Scale (FaCE), and with two disease non-specific instruments, the Hospital Anxiety and Depression Scale (HADS), and Brief-Illness Perception Questionnaire (BIPQ). The efficacy of our clinical intervention will be measured with social-perceptual and mental health outcome measurement before and after treatment (AIM 3).

AIM 2: Determine the social, emotional, and functional burden of synkinesis, not captured in current patient-reported outcome measures as well as effect of treatment. Qualitative interviews with individual participants collected before treatment, after four months of treatment, and after eight months of treatment will be analyzed to study the burden of disease, experience with treatment, and potential differences in both treatments. The primary outcome is to identify the domains that may be missing from existing patient-reported measures collected in AIM 1. To do this, findings to assessment domains (i.e. decreased engagement, negative mood, etc.) in the FaCE, SAQ, and the two disease non-specific instruments, HADS and BIPQ will be compared. The investigators will then evaluate their findings based on domains in Patient-Reported Outcomes Measurement Information System (PROMIS) measures, an NIH-supported collection of validated and standardized scales.

AIM 3: Quantify the disruption in social functioning caused by synkinesis using innovative social-perceptual outcomes and emotion recognition tasks. Prior to treatment, participants will enroll in IRB Protocol 2015-0366 and complete a series of social functioning and mental health instruments and emotion expression recognition tasks. Results will be compared to control participants without facial disability to reveal the social-perceptual impairment attributable to synkinesis. Repetition of these tasks after four months of either treatment may show improvement in recognition and emotional information interpretation when compared to initial measurements.

ELIGIBILITY:
Inclusion Criteria:

* Has ipsilateral synkinesis of facial muscles
* It has been at least four months since their onset of peripheral facial paralysis from any cause
* Ability to read and write in English

Exclusion Criteria:

* previous treatment with reanimation surgery (except for upper eyelid weight placement)
* intolerance or contraindication to botulinum toxin injection
* previous treatment for synkinesis with chemodenervation or neuromuscular retraining therapy
* pregnant and/or breastfeeding women
* participants with impaired decision-making capacity, including those with severe psychiatric illnesses

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2019-10-24 (Actual); Primary Completion 2021-08-24 (Actual); Study Completion 2021-08-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Scott R Chaiet, MD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Neuromuscular Retraining Therapy | Chemodenervation
Started | 7 | 8 (8 participants were consented and assigned to this arm; however, 1 never attended clinic visits and therefore no data was collected from or about this participant.)
Completed | 5 | 7
Not Completed | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Neuromuscular Retraining Therapy | Chemodenervation | Total
Number analyzed (Participants) | 7 | 8 | 15
Age, Continuous [Mean (Full Range); unit: years] | 51.57 [42 to 70] | 49.88 [22 to 71] | 50.67 [22 to 71]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 8 | 12
  Male | 3 | 0 | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 7 | 8 | 15
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 6 | 7 | 13
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 7 | 8 | 15
Diagnosis [Count of Participants; unit: Participants]
  Facial nerve paralysis: mixed with Synkinesis | 7 | 7 | 14
  Facial nerve paralysis: Synkinesis only | 0 | 1 | 1
Laterality [Count of Participants; unit: Participants]
  Right | 5 | 5 | 10
  Left | 2 | 3 | 5
Cause of Facial Palsy [Count of Participants; unit: Participants]
  Bell's | 6 | 6 | 12
  Ramsay-Hunt | 0 | 1 | 1
  Trauma | 1 | 0 | 1
  Other | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Change in Sunnybrook Facial Grading System (SFGS) Between Baseline and 4 Month Scoring
Description: Participants will be videotaped as part of routine care and undergo a blinded SFGS scoring. Scoring is determined by a voluntary movement score (5-items scored from 1-5 where 1 is unable to move and 5 is complete voluntary movement - total range of 5-25, multiplied by 4, where a higher score is a better outcome) minus a resting symmetry score (total of 0-4 where 0 is normal and 4 indicates some asymmetry, multiplied by 5, where a lower score is a better outcome) minus a synkinesis score (5-items scored from 0-3 where 0 is none and 3 is severe, a lower score is a better outcome). Total possible range of scores is 20-100, with a higher score being a better outcome. Scores from baseline will be compared to those at 4 months and the change between the two will be reported.
Time Frame: up to 4 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Neuromuscular Retraining Therapy | Chemodenervation
Number analyzed (Participants) | 7 | 7
score on a scale | 0.29 (4.72) | 5.86 (3.72)

2. Secondary Outcome: Synkinesis Assessment Questionnaire (SAQ) at Baseline
Description: The SAQ is a 9-item questionnaire where each item is scored on a scale from 1-5, 1 is seldom or not at all, and 5 is all of the time, or severely. A higher score indicates a worse outcome. The total range in possible scores is 9-100 (summate scores for questions 1-9/45x100 = SAQ total score) with higher scores indicating more severe facial paralysis symptoms. SAQ scores will be collected as part of routine care throughout the study. Scores will be reported for baseline, 4 months (mid-study), and 8 months (end of study).
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Neuromuscular Retraining Therapy | Chemodenervation
Number analyzed (Participants) | 7 | 7
score on a scale | 54.92 (11.67) | 52.70 (23.68)

3. Secondary Outcome: Synkinesis Assessment Questionnaire (SAQ) at 4 Months
Description: as for outcome 2
Time Frame: 4 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Neuromuscular Retraining Therapy | Chemodenervation
Number analyzed (Participants) | 6 | 7
score on a scale | 64.07 (15.55) | 63.18 (16.22)

4. Secondary Outcome: Synkinesis Assessment Questionnaire (SAQ) at 8 Months
Description: as for outcome 2
Time Frame: 8 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Neuromuscular Retraining Therapy | Chemodenervation
Number analyzed (Participants) | 3 | 4
score on a scale | 55.55 (16.02) | 56.67 (26.26)

5. Secondary Outcome: Facial Clinimetric Evaluation Scale (FaCE) at Baseline
Description: The FaCE scale is 15-item self-report survey to assess the symptoms of facial paralysis in the past week. The total possible range of scores is 15-100 where the higher the score, the lesser the symptoms. Scores will be reported for baseline, 4 months (mid-study), and 8 months (end of study).
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Neuromuscular Retraining Therapy | Chemodenervation
Number analyzed (Participants) | 7 | 7
score on a scale | 56.43 (15.85) | 42.14 (25.80)

6. Secondary Outcome: Facial Clinimetric Evaluation Scale (FaCE) at 4 Months
Description: as for outcome 5
Time Frame: 4 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Neuromuscular Retraining Therapy | Chemodenervation
Number analyzed (Participants) | 7 | 7
score on a scale | 63.10 (13.28) | 45.95 (21.45)

7. Secondary Outcome: Facial Clinimetric Evaluation Scale (FaCE) at 8 Months
Description: as for outcome 5
Time Frame: up to 8 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Neuromuscular Retraining Therapy | Chemodenervation
Number analyzed (Participants) | 3 | 4
score on a scale | 71.67 (9.28) | 61.67 (11.63)

8. Secondary Outcome: Hospital Anxiety and Depression Scale (HADS) at Baseline
Description: The HADS instrument measures anxiety and depressive tendency. 7-items are scored for depression with a total score of 0-21 where the higher the score, the more symptoms of depression. 7-items are scored for anxiety with a total score of 0-21 where the higher the score, the more symptoms of anxiety. Scores will be reported for baseline, 4 months (mid-study), and 8 months (end of study).
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Neuromuscular Retraining Therapy | Chemodenervation
Number analyzed (Participants) | 7 | 7
score on a scale
  Anxiety | 6.14 (4.30) | 10.29 (4.15)
  Depression | 5.71 (3.15) | 7.00 (4.47)

9. Secondary Outcome: Hospital Anxiety and Depression Scale (HADS) at 4 Months
Description: as for outcome 8
Time Frame: 4 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Neuromuscular Retraining Therapy | Chemodenervation
Number analyzed (Participants) | 7 | 5
score on a scale
  Anxiety | 6.57 (3.26) | 8.00 (3.74)
  Depression | 4.14 (2.34) | 5.60 (5.13)

10. Secondary Outcome: Hospital Anxiety and Depression Scale (HADS) at 8 Months
Description: as for outcome 8
Time Frame: 8 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Neuromuscular Retraining Therapy | Chemodenervation
Number analyzed (Participants) | 6 | 6
score on a scale
  Anxiety | 6.67 (2.88) | 7.50 (3.67)
  Depression | 5.50 (2.35) | 2.67 (1.75)

11. Secondary Outcome: Brief-Illness Perception Questionnaire (BIPQ) at Baseline
Description: The BIPQ is a 9-item questionnaire, where the first 8-items are scored from 0-10. To determine a composite score, items 3, 4, and 7 should be reversed scored and added to 1, 2, 5, 6, and 8 (total range of possible scores from 0-80). The higher the score the more threatening the illness is perceived to be. Scores will be reported for baseline, 4 months (mid-study), and 8 months (end of study).
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Neuromuscular Retraining Therapy | Chemodenervation
Number analyzed (Participants) | 7 | 7
score on a scale | 40.00 (8.31) | 51.43 (6.45)

12. Secondary Outcome: Brief-Illness Perception Questionnaire (BIPQ) at 4 Months
Description: as for outcome 11
Time Frame: 4 months
Population: 2 participants in the Chemodenervation arm did not progress to 4 months on study and therefore were not analyzed for this measure at this timepoint.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Neuromuscular Retraining Therapy | Chemodenervation
Number analyzed (Participants) | 7 | 5
score on a scale | 31.71 (7.16) | 45.40 (11.17)

13. Secondary Outcome: Brief-Illness Perception Questionnaire (BIPQ) at 8 Months
Description: as for outcome 11
Time Frame: up to 8 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Neuromuscular Retraining Therapy | Chemodenervation
Number analyzed (Participants) | 7 | 6
score on a scale | 32.57 (8.52) | 42.17 (7.52)

14. Secondary Outcome: Pre-Treatment Qualitative Interviews
Description: Qualitative analysis will proceed concurrently with data collection to allow identified themes to be explored in subsequent interviews. In qualitative research this involves both coding the written transcripts and then modeling the coded data. All team members will analyze the data and look for themes and trends that are emergent from the data. For the pre-treatment interviews, Conventional Content Analysis will be employed to obtain direct information from study participants without imposing preconceived categories or theoretical perspectives.
Time Frame: up to 8 months
Population: Data were not collected.
Arm/Group | Neuromuscular Retraining Therapy | Chemodenervation
Number analyzed (Participants) | 0 | 0

15. Secondary Outcome: Post-Treatment Qualitative Interviews
Description: Qualitative analysis will proceed concurrently with data collection to allow identified themes to be explored in subsequent interviews. In qualitative research this involves both coding the written transcripts and then modeling the coded data. All team members will analyze the data and look for themes and trends that are emergent from the data. For post-treatment interviews, directed content analysis will be employed as findings from pre-treatment interviews will guide analysis of post-treatment interviews while capturing emergent themes that come up in the data.
Time Frame: up to 4 months
Measure: Count of Participants; unit: Participants
Arm/Group | Neuromuscular Retraining Therapy | Chemodenervation
Number analyzed (Participants) | 7 | 7
Participants
  Perception of Impact on Life: Improved | 2 | 4
  Perception of Impact on Life: Stayed the same | 4 | 1
  Perception of Impact on Life: Got worse | 1 | 2
  Perception of Impact on Life: Not discussed | 0 | 0
  Perception on Symptom Control: Improved | 6 | 2
  Perception on Symptom Control: Stayed the same | 0 | 4
  Perception on Symptom Control: Got worse | 0 | 1
  Perception on Symptom Control: Not discussed | 1 | 0
  Concern about the disease: Improved | 5 | 2
  Concern about the disease: Stayed the same | 1 | 4
  Concern about the disease: Got worse | 0 | 1
  Concern about the disease: Not discussed | 1 | 0
  Disease Understanding: Improved | 7 | 4
  Disease Understanding: Stayed the same | 0 | 3
  Disease Understanding: Got worse | 0 | 0
  Disease Understanding: Not discussed | 0 | 0
  Perception of Emotional Impact: Improved | 2 | 2
  Perception of Emotional Impact: Stayed the same | 5 | 5
  Perception of Emotional Impact: Got worse | 0 | 0
  Perception of Emotional Impact: Not discussed | 0 | 0
  Overall facial tightness: Improved | 4 | 4
  Overall facial tightness: Stayed the same | 0 | 1
  Overall facial tightness: Got worse | 0 | 0
  Overall facial tightness: Not discussed | 3 | 2
  Tension in forehead: Improved | 1 | 1
  Tension in forehead: Stayed the same | 0 | 0
  Tension in forehead: Got worse | 0 | 0
  Tension in forehead: Not discussed | 6 | 6
  Tightness in cheek: Improved | 3 | 4
  Tightness in cheek: Stayed the same | 3 | 1
  Tightness in cheek: Got worse | 0 | 0
  Tightness in cheek: Not discussed | 1 | 2
  Tightness in mouth: Improved | 4 | 3
  Tightness in mouth: Stayed the same | 3 | 0
  Tightness in mouth: Got worse | 0 | 1
  Tightness in mouth: Not discussed | 0 | 3
  Tightness in neck: Improved | 0 | 3
  Tightness in neck: Stayed the same | 4 | 0
  Tightness in neck: Got worse | 0 | 0
  Tightness in neck: Not discussed | 3 | 4
  Pain from tightness/spasms: Improved | 3 | 4
  Pain from tightness/spasms: Stayed the same | 0 | 0
  Pain from tightness/spasms: Got worse | 0 | 0
  Pain from tightness/spasms: Not discussed | 4 | 3
  Control while eating/drinking: Improved | 6 | 6
  Control while eating/drinking: Stayed the same | 0 | 0
  Control while eating/drinking: Got worse | 0 | 1
  Control while eating/drinking: Not discussed | 1 | 0
  Smile: Improved | 6 | 4
  Smile: Stayed the same | 1 | 3
  Smile: Got worse | 0 | 0
  Smile: Not discussed | 0 | 0
  Enunciation: Improved | 1 | 2
  Enunciation: Stayed the same | 1 | 0
  Enunciation: Got worse | 0 | 1
  Enunciation: Not discussed | 5 | 4
  Other mouth control: Improved | 3 | 5
  Other mouth control: Stayed the same | 2 | 0
  Other mouth control: Got worse | 0 | 1
  Other mouth control: Not discussed | 2 | 1
  Control over eye trigger: Improved | 7 | 4
  Control over eye trigger: Stayed the same | 0 | 1
  Control over eye trigger: Got worse | 0 | 0
  Control over eye trigger: Not discussed | 0 | 2
  Eye closing too much (triggered): Improved | 6 | 5
  Eye closing too much (triggered): Stayed the same | 1 | 0
  Eye closing too much (triggered): Got worse | 0 | 1
  Eye closing too much (triggered): Not discussed | 0 | 1
  Eye closing too much (at rest): Improved | 6 | 2
  Eye closing too much (at rest): Stayed the same | 0 | 1
  Eye closing too much (at rest): Got worse | 1 | 2
  Eye closing too much (at rest): Not discussed | 0 | 2
  Eye watering: Improved | 5 | 2
  Eye watering: Stayed the same | 1 | 3
  Eye watering: Got worse | 0 | 1
  Eye watering: Not discussed | 1 | 1
  General control of muscles: Improved | 4 | 3
  General control of muscles: Stayed the same | 0 | 0
  General control of muscles: Got worse | 0 | 0
  General control of muscles: Not discussed | 3 | 4
  Facial asymmetry: Improved | 4 | 4
  Facial asymmetry: Stayed the same | 0 | 0
  Facial asymmetry: Got worse | 0 | 0
  Facial asymmetry: Not discussed | 3 | 3
  Sounds in ear: Improved | 1 | 0
  Sounds in ear: Stayed the same | 0 | 1
  Sounds in ear: Got worse | 0 | 0
  Sounds in ear: Not discussed | 6 | 6

16. Primary Outcome: Sunnybrook Facial Grading System (SFGS) at Baseline
Description: Participants will be videotaped as part of routine care and undergo a blinded SFGS scoring. Scoring is determined by a voluntary movement score (5-items scored from 1-5 where 1 is unable to move and 5 is complete voluntary movement - total range of 5-25, multiplied by 4, where a higher score is a better outcome) minus a resting symmetry score (total of 0-4 where 0 is normal and 4 indicates some asymmetry, multiplied by 5, where a lower score is a better outcome) minus a synkinesis score (5-items scored from 0-3 where 0 is none and 3 is severe, a lower score is a better outcome). Total possible range of scores is 20-100, with a higher score being a better outcome.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Neuromuscular Retraining Therapy | Chemodenervation
Number analyzed (Participants) | 7 | 7
score on a scale | 65.71 (9.30) | 54.29 (13.21)

17. Primary Outcome: Sunnybrook Facial Grading System (SFGS) at 4 Months
Description: as for outcome 16
Time Frame: 4 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Neuromuscular Retraining Therapy | Chemodenervation
Number analyzed (Participants) | 7 | 7
score on a scale | 66.00 (6.98) | 60.14 (10.90)

18. Primary Outcome: Sunnybrook Facial Grading System (SFGS) at 8 Months
Description: as for outcome 16
Time Frame: 8 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Neuromuscular Retraining Therapy | Chemodenervation
Number analyzed (Participants) | 3 | 4
score on a scale | 73.00 (8.89) | 60.25 (4.03)

ADVERSE EVENTS:
Time Frame: 8 months
Arm/Group | Neuromuscular Retraining Therapy | Chemodenervation
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/8
Other Adverse Events (participants affected / at risk) | 0/7 | 0/8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-04-15): https://cdn.clinicaltrials.gov/large-docs/72/NCT04148872/Prot_SAP_000.pdf